CLINICAL TRIAL: NCT07019415
Title: Effect Supplementation Vitamin D on HbA1c, Insulin, HOMA-IR and VCAM-1 in Diabetes Mellitus Type 2
Brief Title: Efect Supplementation Vitamin D in Diabetes Mellitus Type 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trisakti University (Other)
Responsible Party: Principal Investigator, Pusparini Pusparini, Prof. Dr.dr. Pusparini, Sp.PK, subsp.K.V.(K), Trisakti University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Universitas Trisakti
Record Dates: First submitted 2025-06-04; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Mellitus Type 2 (T2DM)
Keywords: vitamin D supplementation; HbA1c; insulin; HOMA-IR; VCAM-1
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Vitamin D; microcrystalline cellulose; stearic acid; sodium starch glycolate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (Placebo Comparator): this control group received placebo tablet
  Interventions: Drug: Placebo : calcium carbonate 500 mg, microcrystalline cellulose, magnesium stearate, sodium starch glycolate
- vitamin D 5000 IU (Experimental): this group were received vitamin D 5000 IU+placebo
  Interventions: Drug: Vitamin D 5000 IU+ placebo

INTERVENTIONS:
Drug: Vitamin D 5000 IU+ placebo — vitamin D 5000 IU + placebo in the experimental group
  Arms: vitamin D 5000 IU
Drug: Placebo : calcium carbonate 500 mg, microcrystalline cellulose, magnesium stearate, sodium starch glycolate — this placebo group receive placebo tablet ( calcium carbonate 500 mg, microcrystalline cellulose, magnesium stearate, sodium starch glycolate )
  Arms: control group

SUMMARY:
This is double blind randomized controlled trial study using 92 subject with diabetes mellitus type 2divided into 2 group, one group as control and other group as vitamin D group. At the end of study the study subject only left 40 subjects in each group. Vitamin D group received vitamin D 5000 IU and the control group received calcium carbonate, microcrystalline cellulose, magnesium stearate, sodium starch glycolate for 6 months. The goal of this study was to determine whether suplmentation Vitamin D 5000 IU for 6 months have any effect on HbA1c, insulin, HOMA-IR nd VCAM-1 in Diabetes mellitus type 2

DETAILED DESCRIPTION:
Both supplementation tablet were made in the same shape, color, odor and packaging. The study was conducted from August 2024 until March 2025. The inclusion criteria in this study were male and females age 18 - 65 years old, had been diagnosed T2DM, duration T2DM ≤ 3 year, HbA1c > 6,5 %, used single antidibetic, were willing to follow the protocol of the study, and were willing to participate in this study after receiving explanations, by signing informed consent. The exclusion criteria were used insulin therapy, had liver disease, renal, disease, pregnant women, or breast feeding women, alergy, hypercalsemia, had been consuming vitamin D in three months before the study. During the study semiquantitative recording of food frequency was carried out at the beginning of the study, after 3 month and 6 months supplementation.

Subjects who passed the initial screening (age, duration of T2DM, taking one type of oral antidiabetic drug) were subjected to laboratory screening consisting of albumin, SGPT, calcium, creatinine. Furthermore subjects who met the inclusion and exclusion criteria were randomized and examined for blood pressure, pulse rate, body weight, height, abdominal circumference followed by drawing venous blood samples. Blood sampling was performed 3 times, namely at the beginning of the study, after 3 months and 6 months supplementation. Subjects were asked to fast 12 hours before venous blood sampling. A 10 ml venous blood was drawn from each subject, made into serum and frozen at minus 20 degree Celcius for use in the simultaneous determination of fasting blood glucose, HbA1c, vitamin 25(OH)D, fasting insulin, HOMA-IR and VCAM-1 concentrations, after the total number of subjects was reached. In addition albumin, SGPT, calcium and creatinine were also examined to monitor adverse event. The determination of vitamin 25(OH)D was performed by method direct competitive chemiluminescent immunoassay (CLIA), determination of insulin was performed by method sandwich enzyme linked immunosorbent assay .(ELISA), while VCAM-1 was determined by enzyme immunoassay

ELIGIBILITY:
Inclusion Criteria:

* male and females age 18 - 65 years old
* had been diagnosed T2DM,
* duration T2DM ≤ 3 year
* HbA1c > 6,5 %
* used single antidibetic
* were willing to follow the protocol of the study and were willing to participate in this study after receiving explanations, by signing informed consent.

Exclusion Criteria:

* used insulin therapy
* had liver disease, renal disease
* pregnant women, or breast feeding women
* alergy
* hypercalsemia
* had been consuming vitamin D in three months before the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2024-08-06 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Effect of vitamin D supplementation on VCAM-1 | baseline, 3 months and 6 months
  The control and experimental groups were measured at baseline, after 3 months and 6 months vitamin D supplementation on VCAM-1 level
Effect of Vitamin D supplementation on HbA1c | baseline, 3 month and 6 month
  The control and experimental groups were measured at baseline, after 3 months and 6 months vitamin D supplementation on HbA1c level

SECONDARY OUTCOMES:
Effect of supplementation vitamin D on blood fasting insulin | baseline, 3 month, 6 month
  The control and experimental groups were measured at baseline, after 3 months and 6 months vitamin D supplementation on blood fasting insulin
Effect of vitamin D supplementation on HOMA-IR | baseline, 3 month, 6 month
  The control and experimental groups were measured at baseline, after 3 months and 6 months vitamin D supplementation on HOMA-IR

CONTACTS AND LOCATIONS:
Locations (1):
- Trisakti University, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No